CLINICAL TRIAL: NCT07345052
Title: Western Sweden Systemic Sclerosis Project - A Study on Underlying Mechanisms for Disease Development and Predictors of Disease Activity and Treatment Response in Patients With Systemic Sclerosis
Brief Title: Western Sweden Systemic Sclerosis Project
Acronym: WESST
Status: Recruiting | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Yuan Zhang, Researcher, Göteborg University
Other Study IDs: WESST
Record Dates: First submitted 2025-12-15; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Scleroderma, Systemic; Fibrosis; Skin; Fibrosis Lung; Interstitial Lung Disease Due to Systemic Disease
MeSH Terms: conditions — Scleroderma, Systemic; Fibrosis; Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — whole blood for DNA plasma Peripheral blood mononuclear cells (PBMC) skin fibroblasts (subgroup) keratinocytes (subgroup) skin biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy control: Participants do not have diagnosis of systemic sclerosis or other rheumatic diseases.
  Interventions: Other: No Intervention: Observational Cohort
- Participants with SSc: Participants with SSc will be included if they fulfil the American College of Rheumatology (ACR)-European League Against Rheumatism (EULAR) criteria for systemic sclerosis, independently of the time of the diagnosis. Subjects with mixed connective tissue disease will not be included.
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — no intervention

SUMMARY:
The main aim of the project is to identify key-factors involved in the development and progression of Systemic Sclerosis (SSc), a chronic invalidating rheumatic disease characterized by high mortality and insufficient treatment options. A cohort of patients with SSc will be collected at the Sahlgrenska University Hospital in Gothenburg, Skaraborg Hospital in Skövde, and Södra Älvsborg Hospital in Borås (Sweden). Thanks to a holistic approach including integrated analysis of blood, and skin samples as well as DNA, and with the use of state-of-the-art methods, this project aims to identify factors (e.g. genes, proteins, metabolites, and immune cell types) associated with the development of SSc and with the progression to a more aggressive phenotype. Functional studies using in vitro model systems and patient specimens will be also implemented. The findings of the current project could lead to the identification of possible diagnostic and prognostic markers for the disease as well as potential drug targets. This cohort will be also linked to the European Scleroderma Trial and Research (EUSTAR), which is an international SSc research network aiming to coordinate research activities on SSc from groups all over Europe in order to improve treatment, quality of life and mortality of patients with SSc.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with SSc according to the ACR and EULAR classification criteria

Exclusion Criteria:

* Diagnosis of Mixed connective tissue disease
* Not speaking or reading Swedish
* With severe cognitive impairment
* With blood count below specified limits
* Allergy to local anaesthetic (for subjects who will provide a skin biopsy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Data and samples from patients diagnosed with SSc from the Sahlgrenska University Hospital in Gothenburg, Skaraborg Hospital in Skövde, and Södra Älvsborg Hospital in Borås (Sweden) as well as from healthy controls will be collected. The cohort includes 65 participants with SSc and between 27 healthy controls.
  * Participants with SSc will be included if they fulfil the American College of Rheumatology (ACR)-European League Against Rheumatism (EULAR) criteria for systemic sclerosis, independently of the time of the diagnosis11. Participants with mixed connective tissue disease will not be included.
  * Healthy controls will not have diagnosis of systemic sclerosis or other rheumatic disease.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Predictors of disease activity and progression in plasma samples | The analyses will be performed in the entire study cohort at inclusion (including healthy subjects) and at the 2- and 5-year FU for patients with SSc.
  Here we will analyse plasma circulating molecules (including but not limited to metabolites, cytokines, lipids, proteins, antibodies, exosomes etc) to identify factors involved in the pathogenesis of SSc by comparing those factors in plasma from subjects with SSc vs. healthy subjects. We also aim to identify factors involved in the prognosis of SSc by comparing circulating molecules in plasma from subjects with limited form SSc vs. diffuse form SSc. We plan to screen plasma samples from study participants for molecules that can be relevant for the pathogenesis and the prognosis of SSc.

SECONDARY OUTCOMES:
Genetic markers of progression to an aggressive phenotype in subjects with SSc | Baseline DNA
  all DNA samples from our cohort will be subjects to either next generation sequencing or GWAS as well as epigenetic studies. Single nucleotide polymorphisms of interest will also analysed in these specimens. Data will be analysed independently and/or merged with those of other large cohorts from all over Europe to identify genetic factors associated with the development of SSc as well as the prognosis and the response to treatment.
Characterisation of skin cells in relation to SSc pathogenesis and progression | The analyses will be performed in the entire study cohort at inclusion (including healthy subjects) and at the 2- and 5-year FU for patients with SSc.
  Here we will study skin cells involved in the fibrotic processes in the skin, i.e. fibroblasts and keratinocytes, as well as skin immune cells. We aim to define factors that trigger the fibroblasts to switch to a pro-fibrotic phenotype and factors associated with the progression of the skin disease. Fibroblasts, keratinocytes and immune cells will be isolated and cultured from skin biopsies. Metabolomics, lipidomics, and proteomics will be performed on cell extracts. We will also perform functional studies. Single-cell RNA-Seq in skin biopsies will be performed.
Memory B cell compartment and prognosis of SSc | Baseline PBMCs
  The overall aim of this WP is to identify how the memory B cell compartment (CD27dull and/or CD27bright memory B cells) are modulated in patients in the initial phase of SSc, therefore only subjects with onset of Raynaud's phenomenon <5 years will be included, plus up 6 controls. We will determine this by flow cytometry and by immunoglobulin sequencing as well as RNA sequencing in patients during the initial phase of the disease with the goal to find prognostic markers during early disease.
PBMCs subsets and activation in the pathogenesis of SSc. | Baseline, 2- and 5- years FU
  We aim to identify specific subsets of PBMCs associated with pathogenesis of SSc, especially T and B lymphocytes.
Circulating fibrocytes and pathogenesis of SSc. | Baseline, 2- and 5- years FU
  Here we aim to study circulating fibrocytes and to identify factors associated with downregulation of the transition of those cells into myofibroblasts.
Arthritis involvement in SSc. | Baseline, 2- and 5-years follow up
  The aim of this work package is to assess the burden of articular manifestations in systemic sclerosis (SSc) and to develop a validated articular score.
Assessment of Lung Function and Biomarker Profiling in Patients with Systemic Sclerosis through PExA sampling | Up to 2 years
  Patients with systemic sclerosis from the WESST cohort will be invited to undergo PExA sampling.
Assessment of Lung Function in Patients with Systemic Sclerosis through Insert Gas Washout | Up to 2 years
  Patients with systemic sclerosis will undergo insert gas washout.
Assessment of Lung Function in Patients with Systemic Sclerosis through Impulse Oscillometry | Up to 2 years
  Patients with systemic sclerosis will undergo impulse oscillometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Rheumatology clinics, Sahlgrenska University Hospital, Gothenburg, Sweden, Sweden

IPD SHARING:
Plan to Share IPD: Undecided